CLINICAL TRIAL: NCT02746510
Title: Validation of a Clinical Screening Grid for Syndromic Schizophrenia
Acronym: Schizo-CGH-EXM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator departure
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01992-47
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Comparative Genomic Hybridization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Array comparative genomic hybridization (Experimental): The investigators plan to include 150 patients with defined (DSM V) schizophrenia and aged 15 years and more. The clinical grid will be prospectively fulfilled for every patients on the basis of his/her medical history and clinical examination. Array comparative genomic hybridization (CGH-a) will be performed on jugal mucosae sample to detect precisely syndromic forms of schizophrenia linked to the presence of a pathogenic Copy Number Variation (CNV) or a pathogenic sequence variation (exome trio sequencing).
  Interventions: Genetic: Array comparative genomic hybridization

INTERVENTIONS:
Genetic: Array comparative genomic hybridization — For each of the 150 patients deoxyribose nucleic acid (DNA) exactracted from a jugal mucosae sample will be analysed by the cytogeneticist and a CGH-a will be performed.

SUMMARY:
Background:

Nowadays, despite a large number of studies about schizophrenia and genetics, clinical red flags for syndromic forms of schizophrenia remain poorly documented.

DETAILED DESCRIPTION:
Methods: This study aims to validate a short clinical screening grid for syndromic forms of schizophrenia linked to a pathogenic Copy Variation Number (CNV). The investigators plan to include 150 patients with defined (DSM V) schizophrenia and aged 15 years and more. The clinical grid will be prospectively fulfilled for every patients on the basis of his/her medical history and clinical examination. Array comparative genomic hybridization (CGH-a) will be performed on jugal mucosae sample to detect precisely syndromic forms of schizophrenia linked to the presence of a pathogenic Copy Number Variation (CNV).

In subjects with no CNV that may explain the onset of schizophrenia, the investigators would like to complete the investigations with exome trio sequencing. With this type of very clinical approach, the investigators wish to determine which semiological elements should alert the psychiatrists as to the presence of a syndromic form. The objective is to propose at the end of this study a simple and reliable scale, usable in psychiatry consultation, to guide the genetic screening of forms of syndromic schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 15 years and more with a schizophrenia defined by the DSM V criterion
* Informed consent signed by the patient or he/she's legal representant

Exclusion Criteria:

* Pregnancy
* Current psychotic decompensation
* Patient with a known genetic syndrome

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Presence or absence of each criteria from the grid. | During the inclusion visit (45 minutes)
  The following criteria are evaluated:
  Intelectual disability Precocity of the disease (before 15 years) Treatment resistance Confusion Familial history of schizophrenia Visual hallucination Psychomotor regression Pyramidal syndrome Ataxia Dystonia Areflexia Epilepsia Autism spectrum disorder Dysmorphic features ENT or visceral malformation Growth delay

SECONDARY OUTCOMES:
Presence or absence of a pathogenic CNV detected on the CGH-a | 4 months from samples to results
  For each of the 150 patients deoxyribose nucleic acid (DNA) exactracted from a jugal mucosae sample will be analysed by the cytogeneticist and a CGH-a will be performed. The results will be transmited to the principal investigator. The latter will transmit the results to the patients. If necessary a genetic counselling will be provided by a geneticist.
Whole exome sequencing | 6 months
  Searching for mosaic genetic variations that may have occurred secondarily to conception in 30 subjects with ARRAY CGH who do not find any chromosomal imbalance that could explain the symptoms

CONTACTS AND LOCATIONS:
Overall Officials: POISSON Alice, PH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- CH Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No